CLINICAL TRIAL: NCT04183439
Title: A Model of the Relationship Between Technical Error and Adverse Patient Outcome: A Constructive Grounded Theory Study
Brief Title: Modeling Technical Error and Adverse Outcomes
Status: Completed | Type: Observational
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Gary Sutkin, Professor, University of Missouri, Kansas City
Other Study IDs: 17-076
Record Dates: First submitted 2019-11-26; First posted 2019-12-03 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Surgical Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgeons Interviewed: We recruited surgeons from two University academic health centers, one specializing in adults and the other in children. The surgeons were selected through a snowball technique and emailed to participate. DK and GS interviewed eleven surgical attendings representing 10 surgical specialties. (Table 2) Each subject had at least 10 years of experience in their respective fields and regularly taught residents.

SUMMARY:
The investigators' objective was to develop a theoretical model exploring the relationship between technical errors and adverse patient outcomes. To achieve this aim, the investigators interviewed surgeons from a diverse group of surgical specialties, asking them about their adverse outcomes from surgery and their most granular surgical techniques. the investigators' focus was on adverse outcomes that could be predictably associated with imperfect surgical technique and therefore prevented with proper technique.

DETAILED DESCRIPTION:
Background:

Minute technical errors performed by the surgeon have the potential to lead to adverse patient outcomes. The objective was to gain a deeper understanding of this relationship through the development of an intraoperative model.

Materials and Methods:

The investigators used Constructivist Grounded Theory methodology, including a comprehensive review of the literature and interviews with surgeons, focusing on avoidance of technical errors. The investigators used the Observational Clinical Human Reliability Assessment system, which categorizes granular, technical intraoperative errors, as their conceptual framework. The investigators iteratively interviewed surgeons, from multiple adult and pediatric surgical specialties, refined our semi-structured interview, and developed a model. The model remained stable after interviewing 11 surgeons, and it was reviewed it with earlier interviewed surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Surgical teacher

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We recruited surgeons from two University academic health centers, one specializing in adults and the other in children. The surgeons were selected through a snowball technique and emailed to participate. DK and GS interviewed eleven surgical attendings representing 10 surgical specialties. Each subject had at least 10 years of experience in their respective fields and regularly taught residents.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Model of the relationship between minute, technical motions by a surgeon and intraoperative adverse events, and eventually adverse patient outcomes | approximately 2 years
  This is a qualitative study interviewing surgeons about the link between technical motions and adverse patient outcomes. Our primary outcome will be a model, developed from their answers.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Sutkin, Principal Investigator — University Missouri Kansas City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tang B, Hanna GB, Joice P, Cuschieri A. Identification and categorization of technical errors by Observational Clinical Human Reliability Assessment (OCHRA) during laparoscopic cholecystectomy. Arch Surg. 2004 Nov;139(11):1215-20. doi: 10.1001/archsurg.139.11.1215. PMID 15545569